CLINICAL TRIAL: NCT01106079
Title: A Randomised Controlled Trial to Compare Intensive Management vs Standard Care in Early Psoriatic Arthritis
Brief Title: TIght COntrol of Psoriatic Arthritis
Acronym: TICOPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Julia Brown (Other)
Collaborators: Arthritis Research UK (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Julia Brown, Director of CTRU, University of Leeds
Organization: University of Leeds (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR07/8350; 2007-004757-28 (EudraCT Number); 18825 (Other Grant/Funding Number: Arthritis Research UK)
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Psoriatic Arthritis
Keywords: Early psoriatic arthritis; Tight control; Intensive management
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive management (Experimental)
  Interventions: Drug: Intensive management or Tight control
- Standard management (Active Comparator)
  Interventions: Drug: Standard management - Control group

INTERVENTIONS:
Drug: Intensive management or Tight control — Those subjects randomised to the intensive management or tight control arm will be reviewed every 4 weeks (by the Principal Investigator at each site or a designated researcher) and will be treated according to a rapidly escalating regime, involving standard DMARDs and biologics. Initial therapy will be with oral methotrexate, increasing in dose rapidly over the first 8 weeks of the study. From the 12 week visit onwards, escalation of therapy in this arm will be performed if subjects do not meet the objective target of Minimal Disease Activity. Initial escalation will be to combination DMARD therapy. If patients in the tight control arm fail to meet the MDA criteria and fulfil the NICE criteria for the use of TNF blockers in psoriatic arthritis at 24 weeks, then they will be offered treatment with these medications. Therapy will continue to be modified throughout the 48 week follow-up until a state of minimal disease activity is reached.
  Arms: Intensive management
Drug: Standard management - Control group — The control group will be seen every 12 weeks in a general rheumatology clinic and will receive standard care, involving standard DMARDs and biologics as appropriate. Treatment will be prescribed as felt appropriate by the treating physicians with no set protocol and no restrictions.
  Arms: Standard management

SUMMARY:
The purpose of this study is to investigate whether tight control of patients with newly diagnosed psoriatic arthritis (consisting of regular 4 weekly objective assessment of disease activity and protocol-led intensive treatment) can improve outcome as opposed to standard care (usually 3 monthly reviews with no objective outcome measures and no protocol for treatment). The principle hypothesis of this study is that tight control of inflammation in psoriatic arthritis using a treatment protocol and pre-defined objective targets for treatment will lead to an improvement in patients' disease activity and a reduction in radiological joint damage.

DETAILED DESCRIPTION:
The TICOPA trial is designed as a randomised, controlled, parallel group, open label, multi-centre clinical trial of 206 patients with recent onset psoriatic arthritis. Patients will be randomised on a 1:1 basis to receive either standard care (12 weekly review) or tight control (4 weekly review) for a period of 48 weeks. The hypothesis is that tight control of inflammation will lead to a better outcome in terms of joint inflammation, joint damage, pain and quality of life for people with PsA. This imaging undertaken within the study will provide a further measure of joint inflammation and damage and will improve understanding of the relationships between inflammation, damage and bony proliferation in psoriatic arthritis.

Those subjects randomised to the tight control arm will be reviewed every 4 weeks (by the PI at each site or a designated researcher), and will be treated according to a rapidly escalating regime, involving standard DMARDs and biologics. Initial therapy will be with oral methotrexate, increasing in dose rapidly over the first 8 weeks of the study. From the 12 week visit onwards, escalation of therapy in this arm will be performed if subjects do not meet the objective target of Minimal Disease Activity. Initial escalation will be to combination DMARD therapy. If patients in the tight control arm fail to meet the MDA criteria and fulfil the NICE criteria for the use of TNF blockers in psoriatic arthritis at 24 weeks, then they will be offered treatment with these medications. Therapy will continue to be modified throughout the 48 week follow-up until a state of minimal disease activity is reached. The control group will be seen every 12 weeks in a general rheumatology clinic and will receive standard care, involving standard DMARDs and biologics as appropriate. Treatment will be prescribed as felt appropriate by the treating physicians with no set protocol and no restrictions.

All subjects will be treated and followed-up for 48 weeks from randomisation according to their treatment allocation and will have 12 weekly clinical disease assessments throughout this period by a fully trained, blinded assessor. This will include measures of disease activity in all of the five aspects of PsA (joint disease, skin disease, enthesitis, dactylitis and spinal disease).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of psoriatic arthritis by a consultant Rheumatologist with less than 24 months disease duration.
* Active disease defined by at least one tender or swollen joint or active enthesitis.
* Age ≥18 years at the time of signing the informed consent form and either male or female patients.
* Patient understands the objectives of the study and is able and willing to sign the Informed Consent Form.
* Men and women of child bearing potential (WCBP) must use at least one adequate birth control measure for the duration of the study and should continue such precautions for 6 months after receiving the last dose of protocol treatment.
* Adequate full blood count within 28 days before randomisation:

  * Haemoglobin count > 8.5 g/dL
  * White blood count (WBC) > 3.5 x 10*9/L
  * Absolute neutrophil count (ANC) > 1.5 x 10*9/L
  * Platelet count > 100 x 10*9/L
* Adequate hepatobiliary function within 28 days before randomisation:

  *ALT and/or AST levels must be within 3 times the upper limit of normal range (ULN) for the laboratory conducting the test.
* The patient must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Previous treatment for articular disease with disease modifying drugs (DMARDs) including, but not limited to, methotrexate, sulfasalazine, leflunomide,
* Women who are pregnant, lactating or planning pregnancy within 6 months of their last dose of protocol treatment.
* Use of any investigational agents within 4 weeks or within 5 half-lives of the investigational agent, whichever is longer, prior to randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving an ACR20 response. | 48 weeks
  To compare intensive management with standard care in terms of the proportion of patients achieving an ACR20 response at 48 weeks post-randomisation, in order to determine whether intensive management has superior clinical efficacy.

SECONDARY OUTCOMES:
Additional clinical efficacy outcomes | 24 weeks
  To compare intensive management with standard care in terms of additional clinical efficacy outcomes at 24 and 48 weeks, including:
  * ACR20 (24 weeks), ACR50 and ACR70
  * PASI 20, PASI 75 and PASI 90
  * Change in Sharp-van der Heijde Score
  * ASAS 20 and ASAS 40
  * Change in enthesitis score
  * Change in dactylitis score
  * Change in mNAPSI
  * Change in HAQ
  * Change in other scores (including BASDAI, tender and swollen joint counts, patient and clinician VAS scores)
  * MDA score
Comparison between intensive management and standard care in terms of Quality of Life (QoL),using PsAQoL | 24 weeks
  To compare intensive management with standard care in terms of Quality of Life (QoL),using PsAQoL between intensive management and standard care at baseline, 24 and 48 weeks
To compare intensive management with standard care in terms of cost effectiveness | 12 weeks
  To compare intensive management with standard care in terms of cost effectiveness at 12, 24 and 48 weeks
Number of participants with adverse events as a measure of safety and tolerability | From baseline until 52 weeks
  To compare intensive management with standard care in terms of safety outcomes over the course of the treatment until 52 weeks
Imaging efficacy: PsAMRIS and ultrasound assessment of disease | 48 weeks
  To compare intensive management with standard care in terms of imaging efficacy outcomes including change in Psoriatic Arthritis Magnetic Resonance Imaging Score (PsAMRIS) and ultrasound assessment of disease at 48 weeks in order to assess inflammation and damage.
Additional clinical efficacy outcomes | 48 weeks
  To compare intensive management with standard care in terms of additional clinical efficacy outcomes at 24 and 48 weeks, including:
  * ACR20 (24 weeks), ACR50 and ACR70
  * PASI 20, PASI 75 and PASI 90
  * Change in Sharp-van der Heijde Score
  * ASAS 20 and ASAS 40
  * Change in enthesitis score
  * Change in dactylitis score
  * Change in mNAPSI
  * Change in HAQ
  * Change in other scores (including BASDAI, tender and swollen joint counts, patient and clinician VAS scores)
  * MDA score
Comparison between intensive management and standard care in terms of Quality of Life (QoL),using PsAQoL | 48 weeks
  To compare intensive management with standard care in terms of Quality of Life (QoL),using PsAQoL between intensive management and standard care at baseline, 24 and 48 weeks.
To compare intensive management with standard care in terms of cost effectiveness | 24 weeks
  To compare intensive management with standard care in terms of cost effectiveness at 12, 24 and 48 weeks
To compare intensive management with standard care in terms of cost effectiveness | 48 weeks
  To compare intensive management with standard care in terms of cost effectiveness at 12, 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Helliwell, Principal Investigator — University of Leeds
Locations (3):
- United Kingdom (3):
  - Chapel Allerton Hospital, Leeds, West Yorkshire
  - St Luke's Hospital, Bradford
  - York District Hospital, York

REFERENCES:
- [Derived] Coates LC, Mahmood F, Emery P, Conaghan PG, Helliwell PS. The dynamics of response as measured by multiple composite outcome tools in the TIght COntrol of inflammation in early Psoriatic Arthritis (TICOPA) trial. Ann Rheum Dis. 2017 Oct;76(10):1688-1692. doi: 10.1136/annrheumdis-2017-211137. Epub 2017 Jun 12. PMID 28606970
- [Derived] O'Dwyer JL, Meads DM, Hulme CT, Mcparland L, Brown S, Coates LC, Moverley AR, Emery P, Conaghan PG, Helliwell PS. Cost-Effectiveness of Tight Control of Inflammation in Early Psoriatic Arthritis: Economic Analysis of a Multicenter Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Mar;70(3):462-468. doi: 10.1002/acr.23293. Epub 2018 Jan 30. PMID 28544822
- [Derived] Coates LC, Moverley AR, McParland L, Brown S, Navarro-Coy N, O'Dwyer JL, Meads DM, Emery P, Conaghan PG, Helliwell PS. Effect of tight control of inflammation in early psoriatic arthritis (TICOPA): a UK multicentre, open-label, randomised controlled trial. Lancet. 2015 Dec 19;386(10012):2489-98. doi: 10.1016/S0140-6736(15)00347-5. Epub 2015 Oct 1. PMID 26433318
- [Derived] Freeston JE, Coates LC, Nam JL, Moverley AR, Hensor EM, Wakefield RJ, Emery P, Helliwell PS, Conaghan PG. Is there subclinical synovitis in early psoriatic arthritis? A clinical comparison with gray-scale and power Doppler ultrasound. Arthritis Care Res (Hoboken). 2014 Mar;66(3):432-9. doi: 10.1002/acr.22158. PMID 24022986
- [Derived] Coates LC, Navarro-Coy N, Brown SR, Brown S, McParland L, Collier H, Skinner E, Law J, Moverley A, Pavitt S, Hulme C, Emery P, Conaghan PG, Helliwell PS. The TICOPA protocol (TIght COntrol of Psoriatic Arthritis): a randomised controlled trial to compare intensive management versus standard care in early psoriatic arthritis. BMC Musculoskelet Disord. 2013 Mar 21;14:101. doi: 10.1186/1471-2474-14-101. PMID 23517506